CLINICAL TRIAL: NCT02426281
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Nab-pacliatxel Plus Gemcitabine in Korean Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Nab-pacliatxel Plus Gemcitabine in Korean Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joon Oh Park, Samsung Medical Center, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-10-061
Record Dates: First submitted 2015-04-15; First posted 2015-04-24 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nab-paclitaxel in combination with gemcitabine (Experimental): nab-paclitaxel in combination with gemcitabine nab- paclitaxel 125mg/m2 in combination with gemcitabine 1000mg/m2 D1, 8 15 every 4 weeks.
  Interventions: Drug: nab-paclitaxel; Drug: gemcitabine

INTERVENTIONS:
Drug: nab-paclitaxel — nab- paclitaxel 125mg/m2 D1, 8 15 every 4 weeks.
  Other Names: ABRAXANE; ABI-007
Drug: gemcitabine — gemcitabine 1000mg/m2 D1, 8 15 every 4 weeks.

SUMMARY:
Nab-paclitaxel (interchangeable with ABRAXANE and ABI-007) is a unique protein formulation of a noncrystalline, amorphous form of paclitaxel in an insoluble particle state. Nab-paclitaxel was designed to improve the chemotherapeutic effects of paclitaxel by exploiting endogenous transport pathways to deliver higher doses of paclitaxel to the tumor and to reduce the solvent-related hypersensitivity and other toxicities associated with Taxol® (paclitaxel) injections, the solvent Cremophor EL, and ethanol vehicle. Nab-paclitaxel provides more rapid tissue distribution and increased tumor accumulation compared to cremophor-EL paclitaxel. Mechanistically, albumin receptor-mediated transport across the endothelium, binding to interstitial proteins, and macropinocytic or receptor-mediated uptake into tumor cells as well as sequestration of paclitaxel by cremophor-EL may contribute to the observed differences. Furthermore, nab-paclitaxel synergizes with gemcitabine in preclinical models. The Cremophor EL-free medium enables nab-paclitaxel to be given at a higher dose and in a shorter duration without the need for premedication to prevent solvent-related hypersensitivity reactions. As of March 2014, nab-paclitaxel is approved under the trade name of ABRAXANE in over 45 countries/regions, including the US, Canada, India, European Union/European Economic Area, South Korea, China, Australia, Bhutan, United Arab Emirates, Nepal, New Zealand, Japan, Russia, Sri Lanka, Argentina, Hong Kong, and Lebanon for the treatment of patients with metastatic breast cancer. ABRAXANE is also approved for the first-line treatment of locally advanced or metastatic non small cell lung cancer (NSCLC) in the US, Japan, Argentina, Australia, and New Zealand, for treatment of advanced gastric cancer in Japan, and for first-line treatment of metastatic adenocarcinoma of the pancreas in the US, EU/EEA, Australia, New Zealand and Argentina.

DETAILED DESCRIPTION:
Preclinical studies have demonstrated that nab-paclitaxel may play a role in sensitizing the tumor to chemotherapeutic agents and specifically increases the antitumor efficacy when combined with gemcitabine. While the mechanism of action for the synergy is unclear, preclinical studies have generated hypothetical models. One hypothesis is a remodeling and weakening of the stroma barrier, allowing the chemotherapeutic agents to have better access to the tumor cells. Weakening the tumor-stroma barrier is particularly important in cancer that is characterized by dense stroma, such as pancreatic cancer. In mice with primary patient derived pancreatic tumor xenografts, nab-paclitaxel plus gemcitabine versus gemcitabine alone resulted in increased tumor regression and depleted the desmoplastic stroma as observed by the less dense, disorganized, wisps of collagen type1 fibers after 4 weeks of treatment. In this study, the intratumoral concentration of gemcitabine was increased by 2.8-fold after 5 days of treatment when nab-paclitaxel was added to gemcitabine. It was hypothesized that nab-paclitaxel may play a role in reducing the dense stroma and may have contributed to the increased intratumoral gemcitabine uptake. Additional preclinical studies in a genetically engineered mouse model of pancreatic adenocarcinoma, coadministration of nab-paclitaxel and gemcitabine also demonstrated tumor regression and increased intratumoral gemcitabine levels after 8 days of treatment. Apoptosis of tumor epithelial cells were observed; however, there were no changes in stromal components or collagen density in this short term treatment model. The increased intratumoral gemcitabine levels were attributed to a marked decrease in the primary gemcitabine metabolizing enzyme, cytidine deaminase, by nab-paclitaxel. Finally, a recent clinical study in subjects with resectable pancreatic cancer treated with neoadjuvant nab-paclitaxel plus gemcitabine showed reduction in fibrotic collagenous stroma, further supporting a stroma active mechanism for nab-paclitaxel.

In a clinical Phase 1/2 dose ranging study (CA040, NCT003980860), nab-paclitaxel plus gemcitabine (CA040, NCT003980860) antitumor activity and tolerability were established in patients who had no prior treatment for metastatic pancreatic cancer. The maximum tolerated dose and recommended dose for further studies was determined to be 125 mg/m2 nab-paclitaxel in combination with 1000 mg/m2 gemcitabine.

In the subsequent randomized international Phase 3 study (MPACT, CA046, NCT00394251) that enrolled 861 patients with metastatic pancreatic cancer, nab-paclitaxel in combination with gemcitabine exhibited a clinically meaningful, statistically significant improvement in OS and progression-free survival (PFS). The median OS (primary endpoint) in the intent-to-treat population was 8.5 months (95% CI = 7.89-9.53) with nab-paclitaxel/gemcitabine compared with 6.7 months (95 % CI = 6.01-7.23) with gemcitabine, p < 0.0001, HR = 0.72 (95% CI = 0.617-0.835). Long-term survival was improved in the nab-paclitaxel/gemcitabine arm versus gemcitabine alone, with a 59% increase at 1 year (35% versus 22%) and doubling at 2 years (9% versus 4%). The secondary (PFS, overall response rate [ORR]) and all other efficacy endpoints showed consistent, statistically significant improvements with nab-paclitaxel/gemcitabine, supporting the results from the primary analysis of OS. Specifically, PFS (by independent review) was 5.5 months (95% CI = 4.47-5.95) versus 3.7 months (95% CI = 3.61-4.04) in the nab-paclitaxel/gemcitabine arm versus gemcitabine alone arms, respectively p < 0.0001; HR =0 .69; 95% CI = 0.581-0.821). The improvement in PFS corresponded to a 31% reduction in the risk of progression or death with nab-paclitaxel/gemcitabine. Furthermore, in this study of metastatic unresectable adenocarcinoma of the pancreas, subjects in the combination arm were on therapy longer than those receiving single agent gemcitabine, indicating disease improvement and tolerable treatment. The suitability of the dosing regimen was confirmed by the observation that the majority of patients did not require a dose reduction, and that 71% of nab-paclitaxel doses were delivered at the starting dose of 125 mg/m2. The safety profile for both regimens was consistent with previous reports. Serious life threatening toxicities were not increased; AEs were acceptable and manageable. The most notable differences in toxicity between the 2 treatment arms was peripheral neuropathy, which was cumulative and rapidly reversible with dose delay and reduction, and neutropenia, which was manageable with dose delays and dose reductions. The incremental risks of sepsis and pneumonitis were managed by protocol amendments to increase awareness, and for early diagnosis and treatment to reduce the risk of fatal outcomes. Since the above described initial analysis of the MPACT study, the updated OS with a cutoff of May 2013 showed that the benefit continued to improve with nab-paclitaxel in combination with gemcitabine, with 8.7 versus 6.6 median months, respectively. The updated survival rates also significantly favored nab-paclitaxel plus gemcitabine at year 1 (35% versus 22%), year 2 (10% versus 5%), and year 3 (4% versus 0%) as compared with gemcitabine alone.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma (Islet cell neoplasms or neuroendocrine carcinomas are excluded)
2. ≥ 18 years of age at the time of signing the informed consent document
3. ECOG 0-1
4. At least one measurable lesion according to recist v1.1
5. No prior palliative chemotherapy for the treatment of metastatic pancreatic cancer (Prior treatment with 5-FU or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed if the treatment had been received at least 6 months before enroll).
6. Adequate BM function: ANC ≥1.5 × 109/L; Platelet count ≥100,000/mm2 (100 × 109/L); Hb (Hb) ≥9 g/dL.
7. Adequate liver and renal function (obtained ≤14 days prior to enroll): AST (SGOT), ALT (SGPT) ≤2.5 × upper limit of normal range (ULN), unless liver metastases are clearly present, then ≤5 × ULN is allowed; Total bilirubin 1.5 ≤ ULN; Serum creatinine within normal limits or calculated clearance ≥ 60 mL/min/1.73 m2
8. Albumin level ≥ 3 g/dl
9. Subjects should be asymptomatic for jaundice prior to Cycle 1 Day 1
10. Subject with signed the Informed Consent Form (ICF) prior to participation in any study-related activities.
11. Female of childbearing potential (FCBP) (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [ie, has had menses at any time during the preceding 24 consecutive months]) must:

    * Either commit to true abstinence or agree to the use of 2 physician-approved contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on IP; and for 3 months following the last dose of IP; and
    * Has a negative serum pregnancy test (β-hCG) result at screening
12. Male subjects must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, and for 6 months following IP discontinuation, even if he has undergone a successful vasectomy
13. Subject able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Subject has known symptomatic brain metastases.
2. History of malignancy in the last 5 years.
3. Breast-feeding or pregnant female
4. Patients with plastic biliary stent (Metal biliary stents are allowed.)
5. Subject has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
6. Subject has known historical or active infection with HIV, hepatitis B, or hepatitis C.
7. Subject has undergone major surgery within 4 weeks prior to Cycle 1 Day 1 of treatment in this study.
8. Subject who experienced a recent myocardial infarction, including severe/unstable angina pectoris, coronary/peripheral artery bypass graft, uncontrolled hypertension, clinically significant cardiac dysrhythmia or clinically significant electrocardiogram (ECG) abnormality, significant or uncontrolled cardiovascular disease CHF, and cerebrovascular accident or transient ischemic attack, or seizure disorder in the past year.
9. Subject has a history of allergy or hypersensitivity to any of the study drugs
10. Subjects with history of connective tissue disorders (eg, lupus, scleroderma, arteritis nodosa).
11. Subjects with a history of interstitial lung disease
12. Any other malignancy within 5 years prior to enrollment, with the exception of adequately treated in-situ carcinoma of the prostate (Gleason score ≤ 7), cervix, uteri, or nonmelanomatous skin cancer (all treatment of which should have been completed 6 months prior to enrollment).
13. Patients has > Grade 1 pre-existing peripheral neuropathy (per CTCAE)
14. Subject has serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the subject's safety or the study data integrity.
15. Subject is enrolled in any other clinical protocol or investigational trial with an interventional agent or assessments that may interfere with study procedures.
16. Subject is unwilling or unable to comply with study procedures
17. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 4 months
  The primary endpoint of the study is progression-free survival (PFS) defined as time to progression or death, whichever comes first.

SECONDARY OUTCOMES:
overall survival (OS) | 4 months
  Survival will be measured as the time from the day 1 of first chemotherapy to the date of death.
Response rate | 4 months
  Percentage of response is complete response (CR) or partial response (PR) is defined as the period is maintained.
Disease control rate | 4 months
  Percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents
toxicities (National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0) | 4 months
  Toxicities as measured by Adverse Events(AEs) and Laboratory Results . The severity / intensity of AEs will be graded based upon the subject's symptoms according to the current active minor version of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0)

OTHER OUTCOMES:
Tumor Markers (CA19-9 test) | 4 months
  Tumor Markers as measured by CA19-9 test.
Quality of life questionnaire | 4 months
  Quality of life will be evaluated for nab-paclitaxel in combination with gemcitabine using the EORTC-QLQ-30 and EORTC QLQ- PAN26 questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Joonoh Park, Professor, Study Chair — Samsung Medical Center
Locations (8):
- South Korea (8):
  - Dong-A University Hospital, Busan
  - Gyeongsang National University Hospital, Gyeongsang
  - CHA Bundang Medical Center, Seongnam-si
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei Cancer Center, Seoul